CLINICAL TRIAL: NCT04665167
Title: Feasibility of Online Exposure Therapy and Self-compassion Interventions for Eating and Body Image Concerns Among Young Adult Women
Brief Title: An Intervention for Eating and Body Image Concerns Among Young Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 168743
Record Dates: First submitted 2020-11-23; First posted 2020-12-11 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-08

CONDITIONS: Eating Disorder Symptom; Body Image Disturbance
Keywords: eating pathology; body image; exposure; self-compassion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body image exposure (Active Comparator): Guided non-judgmental exposure, 40 minutes total
  Interventions: Behavioral: Body image exposure
- Self-compassion (Active Comparator): 8 Short self-compassion meditations, 40 minutes total
  Interventions: Behavioral: Self-compassion

INTERVENTIONS:
Behavioral: Body image exposure — Exposure therapy is a key element of evidence-based cognitive behaviour therapy for eating disorders . Body image exposure intervention involves deliberate, planned, and systematic exposure to the body image. Participants will be asked to stand so that they can see their whole body - far enough back. Participants will be asked to look at their bodies on screen. Participants will be continually encouraged by the facilitator for looking at and talking about the body parts.
  Arms: Body image exposure
Behavioral: Self-compassion — The self-compassion intervention condition consists of Neff's self-compassion exercises. These exercises are part of the self-compassion intervention condition. Meditation text used in this study is obtained from the following link https://self-compassion.org/category/exercises/.
  Arms: Self-compassion

SUMMARY:
The primary aim of the current study is to assess acceptability and feasibility of online body image exposure and self-compassion interventions before conducting a larger RCT.

DETAILED DESCRIPTION:
This study will determine the feasibility and effectiveness of delivering an online therapy for eating pathology and body image disturbance. It will address body image and eating pathology in a non-clinical group of young adult women, who are at risk of developing such problems . The feasibility study will determine whether there are any difficulties that would need to be addressed in recruitment, online delivery and assessment of those treatments.

ELIGIBILITY:
Inclusion Criteria:

* Body shape questionnaire score > 25
* Age ≥18
* Self-identified women
* Be able to use a computer and having an Internet connection and webcam

Exclusion Criteria:

* Insufficient knowledge of English
* Learning disability, severe mental illness or alcohol/substance dependence, history of self-injuries, current eating disorder, current clinical depression
* Psychiatric illness requiring secondary care intervention
* Male
* Under 18 years old
* Body mass index below 18.5
* Currently undergoing psychological therapies
* No access to a tablet or computer with an internet connection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified women
Enrollment: 30 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited | will measure upon study termination (estimated at 2-3 months)
  30 participants

SECONDARY OUTCOMES:
The rate of completion | will measure upon study termination (estimated at 2-3 months)
  assessed by the percentage of participants who complete the study questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Fidan Turk, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, United Kingdom

REFERENCES:
- [Background] Franko DL, Striegel-Moore RH. The role of body dissatisfaction as a risk factor for depression in adolescent girls: are the differences Black and White? J Psychosom Res. 2002 Nov;53(5):975-83. doi: 10.1016/s0022-3999(02)00490-7. PMID 12445587
- See also: NICE, 2017. Eating disorders: recognition and treatment — http://www.nice.org.uk/guidance/ng69/resources/eating-disorders-recognition-and-treatment-pdf-1837582159813